CLINICAL TRIAL: NCT03912428
Title: Evaluation of a Novel PET Radioligand as an Inflammatory Biomarker in Musculoskeletal Conditions
Brief Title: Novel PET Radioligand as an Inflammatory Biomarker in Musculoskeletal Conditions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to difficulty with participant recruitment and data futility
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 190079; 19-M-0079
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Myositis; Inflammatory; Rheumatoid Arthritis; Healthy Volunteers
Keywords: Inflammatory; PET Imaging
MeSH Terms: conditions — Myositis; Arthritis, Rheumatoid | interventions — (11C)-MC1; Celecoxib; Positron-Emission Tomography; Radionuclide Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Pilot - Whole body scan in health participants (Other): Healthy participants receive about 10 mCi of [11C]MC1 intravenously followed by a whole body PET/CT scan. If radiation dose to selected body organs is within safety limit, Phase 2 of study was initiated
  Interventions: Drug: 11C-MC1; Diagnostic Test: Positron Emission Tomography (PET)/computed tomography (CT) Scan
- Phase 2: Whole body PET/CT scans in patients (Other): Participants with rheumatoid arthritis (RA), idiopathic inflammatory myopathies (IIM), or axial spondyloarthritis (AXSPA), had a baseline whole body PET/CT scan after about 15 mCi of [11C]MC1 followed by a second whole body PET/CT scan with about 15 mCi of [11C]MC1 intravenously after blockade with single dose of celecoxib 200-400 mg orally on same day.
  Interventions: Drug: 11C-MC1; Drug: Celecoxib; Diagnostic Test: Positron Emission Tomography (PET)/computed tomography (CT) Scan
- Phase 2: Whole body PET/CT scans in healthy participants (Other): Healthy participants had a baseline whole body PET/CT scan after receiving about 15 mCi of [11C]MC1 followed by a second whole body PET/CT scan with about 15 mCi of [11C]MC1 intravenously after blockade with single dose of celecoxib 200-400 mg orally on same day. In a second visit, participants had a baseline whole body PET/CT scan after receiving about 15 mCi of [11C]ER176 followed by a second whole body PET/CT scan with about 15 mCi of [11C]ER176 intravenously after blockade with single dose of celecoxib 200-400 mg orally on same day.
  Interventions: Drug: 11C-MC1; Drug: Celecoxib; Drug: [11C]ER176; Diagnostic Test: Positron Emission Tomography (PET)/computed tomography (CT) Scan
- Phase 3: Brain PET/CT scans in healthy participants (Other): Healthy participants had a baseline brain PET/CT scan after receiving about 20 mCi [11C]MC1 followed by a second brain PET/CT scan with 20 mCi [11C]MC1 intravenously after blockade with single dose of celecoxib 600 mg orally on same day. Participants had arterial blood sampling with each brain scan.
  Interventions: Drug: 11C-MC1; Drug: Celecoxib; Diagnostic Test: Positron Emission Tomography (PET)/computed tomography (CT) Scan

INTERVENTIONS:
Drug: 11C-MC1 — PET radioligand for Cyclooxygenase-2 (COX-2)
Drug: Celecoxib — Cyclooxygenase-2 (COX-2) inhibitor
  Other Names: Celebrex
  Arms: Phase 2: Whole body PET/CT scans in healthy participants; Phase 2: Whole body PET/CT scans in patients; Phase 3: Brain PET/CT scans in healthy participants
Drug: [11C]ER176 — Radioligand for 18-kDa Translocator Protein
  Arms: Phase 2: Whole body PET/CT scans in healthy participants
Diagnostic Test: Positron Emission Tomography (PET)/computed tomography (CT) Scan — Whole body or brain PET/CT scans

SUMMARY:
Background:

Inflammation plays a significant role in various disorders that involve neurodegeneration or autoimmune reaction as one of their mechanisms. PET scans can help detect inflammation. Two new drugs may create better PET images.

Objective:

- To see if the drug [11C]MC1 can help image inflammation.

Eligibility:

* People age 18 and older with rheumatoid arthritis or idiopathic inflammatory myopathy (IIM).
* Healthy volunteers enrolled in protocol 01-M-0254 or 17-M-0181 are also needed.

Design:

* Healthy participants will be screened under protocol 01-M-0254 or 17-M-0181.
* Participants with arthritis or IIM will have a screening visit. This will include:
* Medical history
* Physical exam
* Blood and urine tests
* Possible CT or X-ray: A machine will take pictures of the body.
* Healthy participants will have 1 or 2 visits. They may have urine tests. They may take the drug celecoxib by mouth. They will have a PET scan. A small amount of one or both study drugs will be injected through a catheter: A needle will guide a thin plastic tube into an arm vein. Another catheter will draw blood. They will like on a bed that slides into a machine. Their vital signs and heart activity will be measured.
* Participants with arthritis will have up to 2 visits after screening. They may take celecoxib and have PET scans.
* Participants with IIM will have up to 3 visits after screening. At 1 or 2 visits, they will take celecoxib and have PET scans. They will have 1 visit where they have an MRI: They will lie on a table that slides into a machine. The machine takes pictures of the body.

DETAILED DESCRIPTION:
I. Objective

18-kDa translocator protein (TSPO) and cyclooxygenase-2 (COX-2) are both implicated in the pathophysiology of various inflammatory disorders, suggesting that both may serve as potential biomarkers of inflammation in brain as well as periphery. Our laboratory recently developed two new radioligands: [11C]ER176 to image TSPO and [11C]MC1 to image COX-2. Using wholebody imaging, this study seeks to determine whether PET imaging using these new radioligands can differentiate two inflammatory conditions-rheumatoid arthritis (RA) and idiopathic inflammatory myopathies (IIM)-from healthy conditions. To determine if [11C]MC1 uptake is specific to COX-2, we will also conduct a blocking study with a selective COX-2 inhibitor (celecoxib) in both [11C]MC1 and [11C]ER176 scans; celecoxib is expected to block uptake of [11C]MC1 but not [11C]ER176. Using brain-dedicated imaging, this seeks to determine whether RA patients and healthy volunteers have specific binding in brain - i.e., uptake that can be blocked celecoxib.

II. Study population

Healthy volunteers (n = 17), patients with RA (n = 15), and patients with IIM (n = 15) will undergo whole-body PET/CT scans. Patients with AxSpA (n=15) will undergo two whole-body PET/MRI scans. In addition, healthy volunteers (n = 22) and patients with RA (n = 12) will have brain-dedicated imaging using [11C]MC1 concurrent with arterial blood sampling. Finally, 15 patients with RA will be imaged during a period of moderate to severe symptoms and after clinically indicated treatment for two to four months. Thus, the entire population will be healthy volunteers (n = 39), patients with RA (n = 42), patients with AxSpA (n=15) and patients with

IIM (n = 15).

III. Design

1. Phase 1: We will begin by injecting up to 10 mCi of [11C]MC1 in one healthy male and one healthy female and then conducting a whole body PET scan. Uptake will be measured in the ovaries and testes, and the dose of radioactivity will be calculated. We will proceed only if the dose to these organs with the higher injected activity proposed for Phase 2 will not exceed the limits specified by the Radioactive Drug Research Committee (RDRC).
2. Phase 2: Fifteen RA patients, 15 IIM patients, and 15 age-, sex-, and genotype-matched healthy subjects will undergo two whole-body PET/CT scans using 15 mCi of [11C]ER176 on one day and two whole-body PET/CT scans using 15 mCi of [11C]MC1 on another day. The first scan on each day will serve as the baseline scan for comparison; the second scan on each day will be a blocking study using celecoxib. The [11C]ER176 scans are not mandatory and will be requested at the discretion of the PI.
3. Phase 3: Twelve RA patients and 22 age- and sex-matched healthy subjects will undergo two brain-dedicated PET/CT scans, each using 20 mCi [11C]MC1, and concurrent with arterial blood sampling. The first scan will be a baseline scan, and the second will be after blockade by celecoxib.
4. Phase 4: Fifteen RA patients will be imaged twice with [11C]MC: while having moderate to severe symptoms and after clinically-indicated therapy for about two to four months. Participants will have whole-body scan after injection of 15 mCi of [11C]MC1.

IV. Outcome measures

For whole body imaging, radioligand uptake in a selected region of interest will be quantified as a Standardized Uptake Value (SUV), which normalizes for injected activity and body weight. Possible differences in actual blood radioligand level will be adjusted by venous blood data obtained during the PET scan. Regional uptake after blockade with celecoxib will be expressed as a percentage of the baseline value. The baseline uptake and the percentage blockade by celecoxib of each radioligand will be compared between patients and healthy subjects as well as between inflamed and non-inflamed regions of the body in RA and IIM patients.

For brain-dedicated imaging, the density of COX-2 will be measured with pharmacokinetic modeling and expressed as distribution volume (VT).

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy subjects

* Aged 18 years or older.
* Willing and able to complete all study procedures.
* Able to provide informed consent.
* Healthy based on medical history, physical examination, and laboratory testing.
* Enrolled in protocol 01-M-0254 The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers or 17-M-0181 Recruitment and Characterization of Healthy Research Volunteers for National Institute of Mental Health (NIMH) Intramural Studies.
* Be age and sex-matched with patient groups for the 15 subjects in the Phase 2.

RA patients

* Aged 18 years or older.
* Willing and able to complete all study procedures.
* Able to provide informed consent.
* Have been given a diagnosis of RA based on the published criteria (Aletaha et al., 2010).
* Have moderate to severe symptoms, as defined by a Disease Activity Score in 28 joints with erythrocyte sedimentation rate (DAS28-ESR) score >3.2, but RA patients may be in remission for the repeat scan in phase 4.

IIM patients

* Aged 18 years or older
* Willing and able to complete all study procedures.
* Able to provide informed consent.
* Meets Bohan and Peter criteria ((Bohan and Peter, 1975a, b) for probable or definite dermatomyositis (DM) or polymyositis (PM), or
* Meets criteria for inclusion body myositis (IBM) as defined by Lloyd et al.: 1) finger flexor or quadriceps weakness, and 2) endomysial inflammation, and 3) either invasion of non-necrotic muscle fibers or rimmed vacuoles.

Axial Spondyloarthritis (AxSpA) patients

* Aged 18 years or older.
* Willing and able to complete all study procedures.
* Able to provide informed consent.
* Have been given a diagnosis of AxSpA based on Assessment of Spondylo-Arthritis International Society (ASAS) criteria AxSpA.

EXCLUSION CRITERIA:

1. Common for all participants

   * Because non-steroidal anti-inflammatory drugs (NSAIDs) inhibit COX-2, subjects should not have taken NSAIDs or willow bark tea for two weeks prior to the PET scan.
   * For Phase 2, 3 and 4 *contraindications to taking COX-2 inhibitors that, in the opinion of the investigators, have the potential to affect the results or the safety of the participant.

   These may include:
   * History of hypersensitivity reaction to COX inhibitors or History of aspirin- or NSAID-induced asthma
   * History of upper or lower gastrointestinal bleeding, gastritis, peptic ulcer disease
   * History of uncontrolled gastroesophageal reflux disease (GERD), but not medically controlled GERD
   * Coagulation disorder
   * Thrombocytopenia
   * Glucose-6-phosphate dehydrogenase (G6PD) deficiency
   * History of gout
   * History of hepatic or renal impairment
   * History of cardiovascular disease or presence of cardiovascular risk factors such as uncontrolled or poorly controlled hypertension
   * Current use of probenecid
   * Patients clinically in remission or who have low disease activity

     * Positive HIV infection
     * Any other history of severe medical illness or injury with the potential to affect study data interpretation or to be any medical contraindication to the procedures performed in the study, including active infection and untreated malignancy.
     * Unable to travel to NIH
     * Recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
     * Inability to lie flat on camera bed for at least two hours, including claustrophobia and overweight greater than the maximum for the scanner (500 lb.).
     * Pregnancy or breastfeeding.
     * Participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use affects the function of daily life.
     * NIMH employees or an NIH employee who is a subordinate/relative/co-worker of the investigators.

       * These criteria will not be applied to the two healthy volunteers participating in the Phase 1 of this study*.
2. Healthy subjects

   * Clinically significant laboratory abnormalities based on tests performed under screening protocol 01-M-0254 or 17-M-0181.
3. AxSpA and IIM patients

   * Unable to have an MRI scan (e.g., pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments, metal fragments in the eye).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will also comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule.
Supporting Information: Study Protocol
Time Frame: 18 months after study closure
Access Criteria: De-identified data can be accessed through NIH Biomedical Translational Research Information System (BTRIS)

REFERENCES:
- [Background] Ikawa M, Lohith TG, Shrestha S, Telu S, Zoghbi SS, Castellano S, Taliani S, Da Settimo F, Fujita M, Pike VW, Innis RB; Biomarkers Consortium Radioligand Project Team. 11C-ER176, a Radioligand for 18-kDa Translocator Protein, Has Adequate Sensitivity to Robustly Image All Three Affinity Genotypes in Human Brain. J Nucl Med. 2017 Feb;58(2):320-325. doi: 10.2967/jnumed.116.178996. Epub 2016 Nov 17. PMID 27856631
- [Background] Kreisl WC, Jenko KJ, Hines CS, Lyoo CH, Corona W, Morse CL, Zoghbi SS, Hyde T, Kleinman JE, Pike VW, McMahon FJ, Innis RB; Biomarkers Consortium PET Radioligand Project Team. A genetic polymorphism for translocator protein 18 kDa affects both in vitro and in vivo radioligand binding in human brain to this putative biomarker of neuroinflammation. J Cereb Blood Flow Metab. 2013 Jan;33(1):53-8. doi: 10.1038/jcbfm.2012.131. Epub 2012 Sep 12. PMID 22968319
- [Background] van der Laken CJ, Elzinga EH, Kropholler MA, Molthoff CF, van der Heijden JW, Maruyama K, Boellaard R, Dijkmans BA, Lammertsma AA, Voskuyl AE. Noninvasive imaging of macrophages in rheumatoid synovitis using 11C-(R)-PK11195 and positron emission tomography. Arthritis Rheum. 2008 Nov;58(11):3350-5. doi: 10.1002/art.23955. PMID 18975347
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (first of two parts). N Engl J Med. 1975 Feb 13;292(7):344-7. doi: 10.1056/NEJM197502132920706. No abstract available. PMID 1090839
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (second of two parts). N Engl J Med. 1975 Feb 20;292(8):403-7. doi: 10.1056/NEJM197502202920807. No abstract available. PMID 1089199
- [Derived] Shrestha S, Kim MJ, Eldridge M, Lehmann ML, Frankland M, Liow JS, Yu ZX, Cortes-Salva M, Telu S, Henter ID, Gallagher E, Lee JH, Fredericks JM, Poffenberger C, Tye G, Ruiz-Perdomo Y, Anaya FJ, Montero Santamaria JA, Gladding RL, Zoghbi SS, Fujita M, Katz JD, Pike VW, Innis RB. PET measurement of cyclooxygenase-2 using a novel radioligand: upregulation in primate neuroinflammation and first-in-human study. J Neuroinflammation. 2020 May 2;17(1):140. doi: 10.1186/s12974-020-01804-6. PMID 32359360
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-M-0079.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 participants signed consent
  - One subject withdrew after signing consent and prior to start of study interventions
Groups:
- Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants: Healthy participants receive about 10 mCi of [11C]MC1 intravenously followed by a whole body PET/CT scan. If radiation dose to selected body organs is within safety limit, Phase 2 of study was initiated
Period: Phase 1: Pilot, Dosimetry
Arm/Group | Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants | Phase 2: Whole Body PET/CT Scans in Patients | Phase 2: Whole Body PET/CT Scans in Healthy Participants | Phase 3: Brain PET/CT Scans in Healthy Participants
Started | 2 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2: Whole Body PET/CT Scans
Arm/Group | Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants | Phase 2: Whole Body PET/CT Scans in Patients | Phase 2: Whole Body PET/CT Scans in Healthy Participants | Phase 3: Brain PET/CT Scans in Healthy Participants
Started | 0 | 14 | 2 | 0
Completed | 0 | 9 | 1 | 0
Not Completed | 0 | 5 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 0
Period: Phase 3: Brain PET/CT Scans
Arm/Group | Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants | Phase 2: Whole Body PET/CT Scans in Patients | Phase 2: Whole Body PET/CT Scans in Healthy Participants | Phase 3: Brain PET/CT Scans in Healthy Participants
Started | 0 | 0 | 0 | 12
Completed | 0 | 0 | 0 | 10
Not Completed | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants | Phase 2: Whole Body PET/CT Scans in Patients | Phase 2: Whole Body PET/CT Scans in Healthy Participants | Phase 3: Brain PET/CT Scans in Healthy Participants | Total
Number analyzed (Participants) | 2 | 14 | 2 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 13 | 0 | 12 | 27
  >=65 years | 0 | 1 | 2 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 10 | 1 | 7 | 19
  Male | 1 | 4 | 1 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 0 | 1 | 9
  Not Hispanic or Latino | 2 | 6 | 2 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 0 | 3 | 8
  White | 0 | 4 | 1 | 7 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Uptake of [11C]MC1 by Organs
Description: Participant received whole body PET/CT scan and radioligand uptake of [11C]MC1 in selected body regions of interest was quantified as a Standardized Uptake Value (SUV) using the Siemens Biograph Micro-Computed Tomography (mCT) with an injected dose of 9 mCi. Organ dosimetry was measured as dose per organ in Roentgen Equivalent Man (rem), which is absorbed dose times an organ-specific quality factor.
Time Frame: Up to 120 minutes during each scan
Population: Participants who completed phase 1 of the study.
Measure: Mean (Standard Deviation); unit: (Roentgen Equivalent Man (rem)
Arm/Group | Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants
Number analyzed (Participants) | 2
(Roentgen Equivalent Man (rem)
  Adrenals | 0.11057425 (0.00536093)
  Brain | 0.15445975 (0.00748861)
  Esophagus | 0.06978655 (0.00338344)
  Extrathoracic Tissue | 0.00000000 (0.00000000)
  Gallbladder Wall | 0.54211500 (0.02628316)
  GI-tract: Lower Large Intestine | 0.07955323 (0.00385695)
  Small Intestine | 0.17037900 (0.00826042)
  Stomach | 0.11414533 (0.00553407)
  GI-tract: Upper Large Intestine | 0.17511175 (0.00848988)
  Colon | 0.13402158 (0.00649772)
  Heart Wall | 0.14198250 (0.00688368)
  Kidneys | 0.21555525 (0.01045068)
  Liver | 0.57352325 (0.02780591)
  Lungs | 0.11444650 (0.00554867)
  Lymph Nodes | 0.00000000 (0.00000000)
  Muscle | 0.06802253 (0.00329791)
  Oral Mucosa | 0.00000000 (0.00000000)
  Pancreas | 0.10799275 (0.00523577)
  Red Marrow | 0.19146125 (0.00928254)
  Salivary Glands | 0.00000000 (0.00000000)
  Bone Surfaces | 0.16822775 (0.00815612)
  Skin | 0.05287773 (0.00256365)
  Spleen | 0.08863150 (0.00429709)
  Thymus | 0.06978655 (0.00338344)
  Thyroid | 0.06346188 (0.00307680)
  Urinary Bladder Wall 3 | 0.20565950 (0.00997091)
  Lens | 0.05287773 (0.00256365)
  Effective Dose | 0.14000000 (0.01000000)

2. Primary Outcome: Uptake of [11C]MC1 by Organs - Gender Specific Organs
Description: as for outcome 1
Time Frame: Up to 120 minutes during each scan
Population: Participants who completed phase 1 of the study.
Measure: Number; unit: Roentgen Equivalent Man (rem)
Arm/Group | Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants
Number analyzed (Participants) | 2
Roentgen Equivalent Man (rem)
  Breasts - Female only: number analyzed (Participants) | 1
  Breasts - Female only | 0.05700660
  Ovaries - Female only: number analyzed (Participants) | 1
  Ovaries - Female only | 0.08372325
  Testes - Male only: number analyzed (Participants) | 1
  Testes - Male only | 0.15045450
  Uterus - Female only: number analyzed (Participants) | 1
  Uterus - Female only | 0.08310000

3. Primary Outcome: Phase 2: [11C]MC1 Binding in Inflamed Body Parts - HANDS
Description: The uptake of [11C]MC1 before (baseline) and after blockade by single dose of celecoxib 400mg orally in inflamed regions of the body in patients. The radioligand uptake of [11C]MC1 during whole body PET/CT scans in selected regions of interest was quantified as a Standardized Uptake Value (SUV), which normalizes for injected activity and body weight, using Bruker's PMOD quantification software.
Time Frame: Up to 120 minutes during each scan
Population: Per protocol document, analysis only applies to patients. Data analysis was done on participants who had usable data.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Phase 2: Whole Body PET/CT Scans in Patients
Number analyzed (Participants) | 2
Standard Uptake Value (SUV)
  Baseline | 1.1920415496 (0.29838844946)
  Blocked | 1.190292618 (0.027520757)

4. Primary Outcome: Phase 2: [11C]MC1 Binding in Non-inflamed Body Parts - HANDS
Description: The uptake of [11C]MC1 before (baseline) and after blockade by a single dose of celecoxib 400mg orally in non-inflamed regions of the body in healthy participants. The radioligand uptake of [11C]MC1 during whole body PET/CT scans in selected regions of interest was quantified as a Standardized Uptake Value (SUV), which normalizes for injected activity and body weight, using Bruker's PMOD quantification software.
Time Frame: Up to 120 minutes during each scan
Population: Per protocol document, analysis only applies to healthy participants. Data analysis was done on participants who had usable data.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Phase 2: Whole Body PET/CT Scans in Healthy Participants
Number analyzed (Participants) | 2
Standard Uptake Value (SUV)
  Baseline | 0.07 (0.000509)
  Blocked | 0.13 (0.074459)

5. Primary Outcome: Phase 2: [11C]MC1 Binding in Inflamed Body Parts - KNEES
Description: The uptake of [11C]MC1 before (baseline) and after blockade by a single dose of celecoxib 400mg orally in inflamed regions of the body in patients. The radioligand uptake of [11C]MC1 during whole body PET/CT scans in selected regions of interest was quantified as a Standardized Uptake Value (SUV), which normalizes for injected activity and body weight, using Bruker's PMOD quantification software.
Time Frame: Up to 120 minutes during each scan
Population: Per protocol document, analysis only applies to patients. Data analysis was done on participants who had usable data.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Phase 2: Whole Body PET/CT Scans in Patients
Number analyzed (Participants) | 4
Standard Uptake Value (SUV)
  Baseline | 0.51298372752 (0.071065370092)
  Blocked | 0.565377936 (0.218519988)

6. Primary Outcome: Phase 2: [11C]MC1 Binding Between Non-inflamed Body - KNEES
Description: as for outcome 4
Time Frame: Up to 120 minutes during each scan
Population: Per protocol document, analysis only applies to healthy participants. There was no usable data for analysis as the signal was not detected within the imaging window.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Phase 2: Whole Body PET/CT Scans in Healthy Participants
Number analyzed (Participants) | 2
Standard Uptake Value (SUV)
  Baseline | NA (NA) — There was no usable data for analysis as the signal was not detected within the imaging window.
  Blocked | NA (NA) — There was no usable data for analysis as the signal was not detected within the imaging window.

7. Primary Outcome: Whole Brain Volume of Distribution (VT)/ Free-fraction (fP) of [11C]MC1
Description: The volume of distribution (VT) of [11C]MC1 measured as the brain-to-plasma ratio using the 2-tissue compartmental modeling divided by free-fraction in the plasma of parent radioligand (fP) at baseline and two hours after blockade with single dose of 600 mg celecoxib orally.
Time Frame: Up to 120 minutes during each scan
Population: Participants who completed the PET/CT brain scans in Phase 3 of the study
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Phase 3: Brain PET/CT Scans in Healthy Participants
Number analyzed (Participants) | 10
mL/cm^3
  Baseline | 109 (16)
  Blocked | 81 (12)

ADVERSE EVENTS:
Time Frame: Up to two days after each PET/CT scan visit
Arm/Group | Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants | Phase 2: Whole Body PET/CT Scans in Patients | Phase 2: Whole Body PET/CT Scans in Healthy Participants | Phase 3: Brain PET/CT Scans in Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/14 | 0/2 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/14 | 0/2 | 0/12
Other Adverse Events (participants affected / at risk) | 0/2 | 1/14 | 1/2 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Pilot - Whole Body PET/CT Scan in Health Participants (N=2) | Phase 2: Whole Body PET/CT Scans in Patients (N=14) | Phase 2: Whole Body PET/CT Scans in Healthy Participants (N=2) | Phase 3: Brain PET/CT Scans in Healthy Participants (N=12)
Burning sensation (General disorders) | 0 | 1 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 1
Medical device site pain (General disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Medical device site rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT03912428/Prot_SAP_000.pdf